CLINICAL TRIAL: NCT05390359
Title: Characterization of the Effects on Bioimpedance and the Sensorimotor System After the Application of Percutaneous Electrolysis Protocols on the Patellar Tendon.
Brief Title: Bioimpedance and Sensorimotor Effects of Percutaneous Electrolysis Protocols on the Patellar Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Francisco Ortega Rehabilitacion Avanzada SL (Other)
Collaborators: Ionclinics & DEIONICS. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPTE/2021-BIOZ
Record Dates: First submitted 2022-04-06; First posted 2022-05-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Percutaneous electrolysis; Patellar tendon; Bioimpedance; Sensorimotor system; Percutaneous electrical stimulation

STUDY DESIGN:
Intervention Model Description: Randomized intervention of repeated measures, quadruple-blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The order of the interventions will be randomized by a third person not involved in the treatment, assessment or statistical analysis. Once the care provider has inserted the needle in each subject, the investigator that apply the treatment will choose the treatment protocol assigned on the stimulator, previously programmed and codified. Thus, nobody (participant, care provider, investigator and the outcome assessor) will know what intervention is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-intensity and short-duration (Experimental): The technique consists of the percutaneous electrical stimulation of the tendon applying a galvanic current through a ultrasound-guided needle.
  Interventions: Other: High-intensity and short-duration
- Low-intensity and long-duration (Experimental): The technique consists of the percutaneous electrical stimulation of the tendon applying a galvanic current through a ultrasound-guided needle.
  Interventions: Other: Low-intensity and long-duration
- High-intensity, short-duration and 20 Hz (Experimental): The technique consists of the percutaneous electrical stimulation of the tendon applying a alternating current through a ultrasound-guided needle.
  Interventions: Other: High-intensity, short-duration and 20 Hz
- Sham electrolysis (Sham Comparator): The technique consists of an introduction ultrasound-guided needle without electrical stimulation.
  Interventions: Other: Sham electrolysis

INTERVENTIONS:
Other: High-intensity and short-duration — The ultrasound guided percutaneous electrolysis will be applied in the middle of the patellar tendon.
  The parameters will be 3 squared pulses of a high intensity current (3 mA), that will be applied for 3 seconds with 3 seconds rests between pulses and 1 second of pulses ramp.
  The current will be off on the first 348 seconds of the intervention approximately and the last 18 seconds it will be on. The total treatment time will be 366 seconds.
  Arms: High-intensity and short-duration
Other: Low-intensity and long-duration — The ultrasound guided percutaneous electrolysis will be applied in the middle of the patellar tendon.
  The parameters will be 3 squared pulses of a low intensity direct current (0.1 mA) during 90 seconds, with 3 seconds rests between pulses and 1 second of pulses ramp.
  The total treatment time will be 366 seconds.
  Arms: Low-intensity and long-duration
Other: High-intensity, short-duration and 20 Hz — The ultrasound guided percutaneous electrolysis will be applied in the middle of the patellar tendon.
  The parameters will be 3 pulses of a high intensity compensated biphasic current (3 mA), during 3 seconds with 3 seconds rests between pulses and 1 second of pulses ramp. The alternating frequency will be of 20 Hz and the pulse width of 50 microseconds.
  The current will be off on the first 348 seconds of the intervention approximately and the last 18 seconds it will be on. The total treatment time will be 366 seconds.
  Arms: High-intensity, short-duration and 20 Hz
Other: Sham electrolysis — The control ultrasound guided percutaneous electrolysis will be applied in the middle of the patellar tendon, without electrical stimulation during 366 seconds.
  Arms: Sham electrolysis

SUMMARY:
Percutaneous electrolysis is a physical therapy technique, whose main objective is the treatment of the signs and symptoms associated with tendinopathies by applying a galvanic current through a blunt dry needle. Despite its clinical use being already stablished, the physiological mechanisms underlying this therapy are still unknown and thus, the optimal parameterization. The present study proposes to perform different stimulation protocols of percutaneous electrolysis on healthy subjects patellar tendon to answer those questions.

DETAILED DESCRIPTION:
Intervention will be performed in the middle of the patellar tendon, using ultrasonography to guide the needle insertion, without risk of affecting any adjacent structure. The theoretical basis of the technique is to produce specific controlled changes in the intervened tissue, and the pathological symptoms, through the accumulation of an electric charge. For this reason, the protocols will be the following:

1. High-intensity and short-duration: 3 squared pulses of a high intensity galvanic current (3 mA) for 3 seconds with 3 seconds rests between pulses and 1 second of pulses ramp. The current will be off during the first 348 seconds of the intervention and the last 18 seconds it will be on. The total intervention time will be 366 seconds.
2. Low-intensity and long-duration: 3 squared pulses of a low intensity galvanic current (0.1 mA) during 90 seconds, with 3 seconds rests between pulses and 30 seconds of pulses ramp. The total intervention time will be 366 seconds.
3. High-intensity, short-duration and 20 Hertz (Hz): 3 squared pulses of a high intensity compensated biphasic squared current (3 mA), during 3 seconds with 3 seconds rests between pulses and 1 second of pulses ramp. The alternative frequency of 20 Hz and the pulse width of 50 ms. The current will be off during the first 348 seconds of the intervention and the last 18 seconds it will be on. The total intervention time will be 366 seconds.
4. Sham electrolysis group will got the same intervention, but without applying electrical current.

The study design will be an crossover clinical trial, with randomized order of intervention with repeated measurements. Therefore, each subject will be have the four protocols at randomized order, with a gap of at least one week between them. The study will be full blinded.

The capacity to recruit the inhibitory system will be evaluated by means of conditioned pain modulation. Moreover, somatosensory thresholds will be evaluated in the knee, as well as knee extension strength. In addition, we will undertake continuous measures of the electrical bioimpedance of the patellar tendon, to study the changes produced by the intervention in the different intra and extracellular tissue components.

The conditioned modulation of pain assesment will take place one week before to the intervention, and the remaining measurements will be measured pre-intervention and post-intervention for each protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Between 18 and 45 years old.

Exclusion Criteria:

* to suffer or to have suffered any pathology on the arm on the last 30 days.
* to suffer some disease discouraging current application or needling, as coagulation deficit, etc.
* to suffer some severe disease as diabetes mellitus, cancer, neurology disease, depression, fibromyalgia, etc.
* to suffer some cognitive disorders.
* to consume drugs as coagulants, anti-depressant, pregabalin, neuropeptide, opioids, etc during investigation or the first week before investigation.
* to consume NSAIDS the last 48 hours before investigation or during investigation.
* belonephobia.
* To consume caffeine 2 hours prior to the investigation or perform intense exercise on the same day as the measurement.
* To receive concomitant physical therapy treatments or have previously received percutaneous electrolysis treatment.
* professional athlete
* To be pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Change in pain evoked with Von Frey Filaments. | Pre-intervention and immediately after the intervention
  We will use Von Frey Filaments to apply a 300g pressure in the evaluated areas (tibialis anterior muscle, inferior pole of the patella and patellar tendon). The subject will report the pain intensity verbally administered Numeric rate scale (NRS): 0 will be any pain and 10 will be the maximal perception of pain). The test will be performed with subject's eyes closed.

SECONDARY OUTCOMES:
Change in transcutaneous electrical detection threshold. | Pre-intervention and immediately after the intervention
  We will use a transcutaneous active electrode to evaluate electrical detection threshold on the medial region of the tibia. We will apply an alternating current with a frequency of 2 Hz, a pulse duration of 150 msec and the intensity will be increased progressively. When the subjects perceives the electrical current, the evaluator will record the current intensity as the electrical detection threshold.
Change in percutaneous electrical detection threshold. | Pre-intervention and immediately after the intervention
  We will use the intervention needle as an active electrode to evaluate electrical detection threshold on the patellar tendon. The parameters of the electric current will be 2 Hz and 150 msec of pulse duration and the intensity will be increased progressively. When the subjects perceives the electrical current, the evaluator will record the current intensity as the electrical detection threshold.
Change in pain evoked with a transcutaneous electrical stimulus. | Pre-intervention and immediately after the intervention
  We will use a transcutaneous active electrode to evaluate pain evoked with electrical stimulus on the medial side of the tibia. The parameters of electric current will be 2 hz and 150 msec of pulse duration and the intensity will be x3-4 respect to the electrical detection threshold determined using an electrical transcutaneous stimulus. The subject will report the pain intensity with a verbally administered numeric rate scale (NRS): 0 will be no pain and 10 will be the maximal perception of pain.
Change in pain evoked with a percutaneous electrical stimulus. | Pre-intervention and immediately after the intervention
  We will use the intervention needle as an active electrode to evaluate electrical detection threshold on the patellar tendon. The parameters of electric current will be 2 Hz and 150 msec of pulse duration and the intensity will be x4-6 respect to the electrical detection threshold determined using an electrical percutaneous simulus. The subject will report the pain intensity with a verbally administered numeric rate scale (NRS): 0 will be no pain and 10 will be the maximal perception of pain.
Change in maximum strength during knee extension with dynamometer | Pre-intervention and immediately after the intervention
  The subject will be sitting with 90 degrees knee flexion and the dynamometer located at the ankle. He/she will must extend the knee executing maximal isometric force during 5 seconds, 2 times with 1 minute to rest between them.
Change in surface electromyography signal during knee extension | Pre-intervention and immediately after the intervention
  The subject will be sitting with 90 degrees knee flexion and the dynamometer located at the ankle and a surface electromyography located at the muscles vastus medialis and lateralis, from the muscle quadriceps femoris. He/she will must extend the knee executing maximal isometric force during 5 seconds, 2 times with 1 minute to rest between them.
Questionnaire Victorian Institute of Sport Assessment - Patella (VISA-P) | One week before intervention
  The subject will fulfil the visa-p questionnaire, that assess symptoms, simple test of function, and the ability to play sports, to control that the sample recruited are healthy subjects.
Change in patellar tendon bioimpedance | pre-intervention / baseline, immediately after the introduction the intervention needle and immediately after the intervention
  We will use four needles in the patellar tendon as electrodes to measure bioimpedance with a specific device (ImpediMed´s SFB7). We will measure using 256 frequences ranging from 3 Kilohertz (KHz) to 1 Megahertz (MHz) in different time frames. Firstly, we will measure three times prior to the introduction of the intervention needle. Then we will measure once more after the introduction of the intervention needle. Finally, we will performed four repeated measures after the intervention (immediately, 5, 10 and 15 minutes after of the intervention).
Pain induced during bioimpedance measurement. | Immediately after the intervention, immediately after the introduction the intervention needle and immediately after of the intervention.
  We will continuously measure pain intensity produced by the bioimpedance recording using a digital visual analogue scale (VAS) integrated in a potentiometer: 0 will be no pain and 10 will be the maximal perception of pain.
Conditioned pain modulation | One week before the intervention
  First, we will measure pressure pain threshold with an algometer on the patellar tendon. Then, we will repeat the assesment of the pressure pain threshold on the patellar tendon meanwhile we apply a moderate painful pressure on the contralateral arm (5/10 on a numeric rate scale NRS: 0 will be no pain and 10 will be the maximal perception of pain) with a pressure cuff. The change between both pressure pain threshold will assess the conditioned pain modulation. After, we will repeat the same procedure but using cutaneous electrical threshold instead of pressure.
International Physical Activity Questionnaire (IPAQ) | One week before the intervention
  The subjects will answer International Physical Activity Questionnaire to assess the level of physical activity.
Questionnaire about intervention effects past 24 hours. | 24 hours after the intervention
  The subjects will answer a questionnaire about the intervention effects and the possible side effects.
Pain induced during intervention | During the 16 minutes of intervention
  We will continuously measure pain intensity produced by the intervention using a digital visual analogue scale (VAS) integrated in a potentiometer: 0 will be no pain and 10 will be the maximal perception of pain.
Change in threshold to elicit mechanical perception with Von Frey Filaments | Pre-intervention and immediately after the intervention
  We will use Von Frey Filaments of increasing caliber to apply different pressure forces in the evaluated areas (tibialis anterior muscle, inferior pole of the patella and patellar tendon). The evaluator will score the caliber of the filament that produce a mechanical perception in the subject as the mechanical pressure threshold. The test will be performed with subject's eyes closed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ionclinics & DEIONICS., Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segura León J.M., Medina i Mirapeix F., Valera Garrido F. Adverse effects of percutaneous needle electrolysis in carpal tunnel syndrome. Rev Fisioter Invasiva 2019;2:130
- [Background] Valera Garrido F., Minaya Muñoz F., Ramírez Martínez P., Medina i Mirapeix F. Adverse effects associated to the application of ultrasound-guided percutaneous needle electrolysis. Rev Fisioter Invasiva 2019; 02(02): 115-116.
- [Background] Valera-Garrido, Polidori F, Canet, Botet J, Ramírez F, Calvo P, et al. Clinical criteria for the application of percutaneous needle electrolysis in tendinopathies: An expert Consensus cocument and cross-sectional study among physical therapists. Revista Fisioterapia Invasiva / Journal of Invasive Techniques in Physical Therapy. 2019; 02. 055-061. 10.1055/s-0039-3402789.
- [Result] Abat F, Valles SL, Gelber PE, Polidori F, Jorda A, Garcia-Herreros S, Monllau JC, Sanchez-Ibanez JM. An experimental study of muscular injury repair in a mouse model of notexin-induced lesion with EPI(R) technique. BMC Sports Sci Med Rehabil. 2015 Apr 17;7:7. doi: 10.1186/s13102-015-0002-0. eCollection 2015. PMID 25897404
- [Result] Abat F, Valles SL, Gelber PE, Polidori F, Stitik TP, Garcia-Herreros S, Monllau JC, Sanchez-Ibanez JM. [Molecular repair mechanisms using the Intratissue Percutaneous Electrolysis technique in patellar tendonitis]. Rev Esp Cir Ortop Traumatol. 2014 Jul-Aug;58(4):201-5. doi: 10.1016/j.recot.2014.01.002. Epub 2014 May 10. Spanish. PMID 24821478
- [Result] Abat F, Diesel WJ, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Effectiveness of the Intratissue Percutaneous Electrolysis (EPI(R)) technique and isoinertial eccentric exercise in the treatment of patellar tendinopathy at two years follow-up. Muscles Ligaments Tendons J. 2014 Jul 14;4(2):188-93. eCollection 2014 Apr. PMID 25332934
- [Result] Aparecida da Silva V, Galhardoni R, Teixeira MJ, Ciampi de Andrade D. Not just a matter of pain intensity: Effects of three different conditioning stimuli on conditioned pain modulation effects. Neurophysiol Clin. 2018 Oct;48(5):287-293. doi: 10.1016/j.neucli.2018.06.078. Epub 2018 Jun 25. PMID 29954673
- [Result] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Result] Barlas P, Ting SL, Chesterton LS, Jones PW, Sim J. Effects of intensity of electroacupuncture upon experimental pain in healthy human volunteers: a randomized, double-blind, placebo-controlled study. Pain. 2006 May;122(1-2):81-9. doi: 10.1016/j.pain.2006.01.012. Epub 2006 Mar 9. PMID 16527396
- [Result] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Result] Rees JD, Maffulli N, Cook J. Management of tendinopathy. Am J Sports Med. 2009 Sep;37(9):1855-67. doi: 10.1177/0363546508324283. Epub 2009 Feb 2. PMID 19188560
- [Result] Cardoso TB, Pizzari T, Kinsella R, Hope D, Cook JL. Current trends in tendinopathy management. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):122-140. doi: 10.1016/j.berh.2019.02.001. Epub 2019 Mar 8. PMID 31431267
- [Result] Cannell LJ, Taunton JE, Clement DB, Smith C, Khan KM. A randomised clinical trial of the efficacy of drop squats or leg extension/leg curl exercises to treat clinically diagnosed jumper's knee in athletes: pilot study. Br J Sports Med. 2001 Feb;35(1):60-4. doi: 10.1136/bjsm.35.1.60. PMID 11157465
- [Result] Cook JL, Khan KM, Harcourt PR, Kiss ZS, Fehrmann MW, Griffiths L, Wark JD. Patellar tendon ultrasonography in asymptomatic active athletes reveals hypoechoic regions: a study of 320 tendons. Victorian Institute of Sport Tendon Study Group. Clin J Sport Med. 1998 Apr;8(2):73-7. doi: 10.1097/00042752-199804000-00001. PMID 9641432
- [Result] Cook JL, Malliaras P, De Luca J, Ptasznik R, Morris M. Vascularity and pain in the patellar tendon of adult jumping athletes: a 5 month longitudinal study. Br J Sports Med. 2005 Jul;39(7):458-61; discussion 458-61. doi: 10.1136/bjsm.2004.014530. PMID 15976171
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] de la Cruz Torres B, Albornoz Cabello M, Garcia Bermejo P, Naranjo Orellana J. Autonomic responses to ultrasound-guided percutaneous needle electrolysis of the patellar tendon in healthy male footballers. Acupunct Med. 2016 Aug;34(4):275-9. doi: 10.1136/acupmed-2015-010993. Epub 2016 Jan 20. PMID 26792776
- [Result] Docking SI, Ooi CC, Connell D. Tendinopathy: Is Imaging Telling Us the Entire Story? J Orthop Sports Phys Ther. 2015 Nov;45(11):842-52. doi: 10.2519/jospt.2015.5880. Epub 2015 Sep 21. PMID 26390270
- [Result] Eckenrode BJ, Kietrys DM, Stackhouse SK. PAIN SENSITIVITY IN CHRONIC ACHILLES TENDINOPATHY. Int J Sports Phys Ther. 2019 Dec;14(6):945-956. PMID 31803527
- [Result] Fernandez-Rodriguez T, Fernandez-Rolle A, Truyols-Dominguez S, Benitez-Martinez JC, Casana-Granell J. Prospective Randomized Trial of Electrolysis for Chronic Plantar Heel Pain. Foot Ankle Int. 2018 Sep;39(9):1039-1046. doi: 10.1177/1071100718773998. Epub 2018 May 17. PMID 29771148
- [Result] Figueroa D, Figueroa F, Calvo R. Patellar Tendinopathy: Diagnosis and Treatment. J Am Acad Orthop Surg. 2016 Dec;24(12):e184-e192. doi: 10.5435/JAAOS-D-15-00703. PMID 27855131
- [Result] Fruhstorfer H, Gross W, Selbmann O. von Frey hairs: new materials for a new design. Eur J Pain. 2001;5(3):341-2. doi: 10.1053/eujp.2001.0250. PMID 11558991
- [Result] Goldin M, Malanga GA. Tendinopathy: a review of the pathophysiology and evidence for treatment. Phys Sportsmed. 2013 Sep;41(3):36-49. doi: 10.3810/psm.2013.09.2019. PMID 24113701
- [Result] Golman M, Wright ML, Wong TT, Lynch TS, Ahmad CS, Thomopoulos S, Popkin CA. Rethinking Patellar Tendinopathy and Partial Patellar Tendon Tears: A Novel Classification System. Am J Sports Med. 2020 Feb;48(2):359-369. doi: 10.1177/0363546519894333. Epub 2020 Jan 8. PMID 31913662
- [Result] Hernandez-Sanchez S, Hidalgo MD, Gomez A. Cross-cultural adaptation of VISA-P score for patellar tendinopathy in Spanish population. J Orthop Sports Phys Ther. 2011 Aug;41(8):581-91. doi: 10.2519/jospt.2011.3613. Epub 2011 Jul 12. PMID 21765223
- [Result] Hutchison MK, Houck J, Cuddeford T, Dorociak R, Brumitt J. Prevalence of Patellar Tendinopathy and Patellar Tendon Abnormality in Male Collegiate Basketball Players: A Cross-Sectional Study. J Athl Train. 2019 Sep;54(9):953-958. doi: 10.4085/1062-6050-70-18. Epub 2019 Aug 19. PMID 31424974
- [Result] Jaffrin MY, Morel H. Body fluid volumes measurements by impedance: A review of bioimpedance spectroscopy (BIS) and bioimpedance analysis (BIA) methods. Med Eng Phys. 2008 Dec;30(10):1257-69. doi: 10.1016/j.medengphy.2008.06.009. Epub 2008 Aug 3. PMID 18676172
- [Result] Kregel J, van Wilgen CP, Zwerver J. Pain assessment in patellar tendinopathy using pain pressure threshold algometry: an observational study. Pain Med. 2013 Nov;14(11):1769-75. doi: 10.1111/pme.12178. Epub 2013 Jun 26. PMID 23802873
- [Result] Lopez-Royo MP, Gomez-Trullen EM, Ortiz-Lucas M, Galan-Diaz RM, Bataller-Cervero AV, Al-Boloushi Z, Hamam-Alcober Y, Herrero P. Comparative study of treatment interventions for patellar tendinopathy: a protocol for a randomised controlled trial. BMJ Open. 2020 Feb 16;10(2):e034304. doi: 10.1136/bmjopen-2019-034304. PMID 32066608
- [Result] Maffiuletti NA, Aagaard P, Blazevich AJ, Folland J, Tillin N, Duchateau J. Rate of force development: physiological and methodological considerations. Eur J Appl Physiol. 2016 Jun;116(6):1091-116. doi: 10.1007/s00421-016-3346-6. Epub 2016 Mar 3. PMID 26941023
- [Result] Martin-Pintado-Zugasti A, Rodriguez-Fernandez AL, Fernandez-Carnero J. Postneedling soreness after deep dry needling of a latent myofascial trigger point in the upper trapezius muscle: Characteristics, sex differences and associated factors. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):301-308. doi: 10.3233/BMR-150630. PMID 26406209
- [Result] Moreno C, Mattiussi G, Nunez FJ, Messina G, Rejc E. Intratissue percutaneous electolysis combined with active physical therapy for the treatment of adductor longus enthesopathy-related groin pain: a randomized trial. J Sports Med Phys Fitness. 2017 Oct;57(10):1318-1329. doi: 10.23736/S0022-4707.16.06466-5. Epub 2017 Jan 23. PMID 28116876
- [Result] Muhsen A, Moss P, Gibson W, Walker B, Jacques A, Schug S, Wright A. The Association Between Conditioned Pain Modulation and Manipulation-induced Analgesia in People With Lateral Epicondylalgia. Clin J Pain. 2019 May;35(5):435-442. doi: 10.1097/AJP.0000000000000696. PMID 30801339
- [Result] Rio E, Moseley L, Purdam C, Samiric T, Kidgell D, Pearce AJ, Jaberzadeh S, Cook J. The pain of tendinopathy: physiological or pathophysiological? Sports Med. 2014 Jan;44(1):9-23. doi: 10.1007/s40279-013-0096-z. PMID 24027089
- [Result] Rodriguez-Huguet M, Gongora-Rodriguez J, Rodriguez-Huguet P, Ibanez-Vera AJ, Rodriguez-Almagro D, Martin-Valero R, Diaz-Fernandez A, Lomas-Vega R. Effectiveness of Percutaneous Electrolysis in Supraspinatus Tendinopathy: A Single-Blinded Randomized Controlled Trial. J Clin Med. 2020 Jun 12;9(6):1837. doi: 10.3390/jcm9061837. PMID 32545583
- [Result] Rodriguez-Huguet M, Gongora-Rodriguez J, Lomas-Vega R, Martin-Valero R, Diaz-Fernandez A, Obrero-Gaitan E, Ibanez-Vera AJ, Rodriguez-Almagro D. Percutaneous Electrolysis in the Treatment of Lateral Epicondylalgia: A Single-Blind Randomized Controlled Trial. J Clin Med. 2020 Jul 1;9(7):2068. doi: 10.3390/jcm9072068. PMID 32630241
- [Result] Sdrulla AD, Xu Q, He SQ, Tiwari V, Yang F, Zhang C, Shu B, Shechter R, Raja SN, Wang Y, Dong X, Guan Y. Electrical stimulation of low-threshold afferent fibers induces a prolonged synaptic depression in lamina II dorsal horn neurons to high-threshold afferent inputs in mice. Pain. 2015 Jun;156(6):1008-1017. doi: 10.1097/01.j.pain.0000460353.15460.a3. PMID 25974163
- [Result] Shiose K, Tanabe Y, Ohnishi T, Takahashi H. Effect of regional muscle damage and inflammation following eccentric exercise on electrical resistance and the body composition assessment using bioimpedance spectroscopy. J Physiol Sci. 2019 Nov;69(6):895-901. doi: 10.1007/s12576-019-00702-8. Epub 2019 Aug 6. PMID 31388975
- [Result] Smidt N, van der Windt DA, Assendelft WJ, Mourits AJ, Deville WL, de Winter AF, Bouter LM. Interobserver reproducibility of the assessment of severity of complaints, grip strength, and pressure pain threshold in patients with lateral epicondylitis. Arch Phys Med Rehabil. 2002 Aug;83(8):1145-50. doi: 10.1053/apmr.2002.33728. PMID 12161838
- [Result] Stoychev V, Finestone AS, Kalichman L. Dry Needling as a Treatment Modality for Tendinopathy: a Narrative Review. Curr Rev Musculoskelet Med. 2020 Feb;13(1):133-140. doi: 10.1007/s12178-020-09608-0. PMID 31942676
- [Result] Scott A, Squier K, Alfredson H, Bahr R, Cook JL, Coombes B, de Vos RJ, Fu SN, Grimaldi A, Lewis JS, Maffulli N, Magnusson SP, Malliaras P, Mc Auliffe S, Oei EHG, Purdam CR, Rees JD, Rio EK, Gravare Silbernagel K, Speed C, Weir A, Wolf JM, Akker-Scheek IVD, Vicenzino BT, Zwerver J. ICON 2019: International Scientific Tendinopathy Symposium Consensus: Clinical Terminology. Br J Sports Med. 2020 Mar;54(5):260-262. doi: 10.1136/bjsports-2019-100885. Epub 2019 Aug 9. No abstract available. PMID 31399426
- [Result] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Result] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675